CLINICAL TRIAL: NCT04292938
Title: Ketogenic Diet in McArdle Disease: a Multicentric Single Blind Controlled Trial
Brief Title: McArdle Disease Treatment by Ketogenic Diet
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Collaborators: University of Pisa (Other); University of Messina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 543
Record Dates: First submitted 2020-02-28; First posted 2020-03-03 (Actual); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Glycogen Storage Disease
Keywords: McArdle; Diet; Ketogenic
MeSH Terms: conditions — Glycogen Storage Disease | interventions — Diet, Ketogenic

STUDY DESIGN:
Intervention Model Description: Randomised controlled single blind
Who Masked: Outcomes Assessor
Masking Description: The assessors will be blinded as to the dietary regimen followed by the patient
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketogenic diet (Active Comparator): patients will follow a low carbohydrate high lipid personalized diet causing blood BOHB level to be between 1.5-4 mmol/l for six months
  Interventions: Dietary Supplement: Low carbohydrate ketogenic diet
- control group (No Intervention): Patients will be asked to maintain their usual dietary regimen

INTERVENTIONS:
Dietary Supplement: Low carbohydrate ketogenic diet — Dietary modification, including the use of supplements, with the aim of reaching a lipid/carbohydrate-protein 3:1 ratio with a minimum 1g/Kg/die in protein
  Other Names: Ketogenic
  Arms: Ketogenic diet

SUMMARY:
McArdle's disease or Glycogen storage disease type 5 (GSD5), the most common muscle glycogenosis, is a rare disabling condition with no effective treatment. There are indications that a special dietary regimen could positively influence the disease manifestations. After contradictory indications for protein rich vs carbohydrate rich diets, several preliminary studies and more and more patients own experiences are now pointing to a low carbohydrate ketogenic diet (LCKD) as possibly effective in improving exercise tolerance and reducing muscle damage. The investigators propose a multicentre randomized single blind controlled trial testing efficacy of an individualized LCKD in GSD5. The investigators will test the ability of a 6 months dietary regimen with a 3:1 LCKD inducing a BOHB blood concentration of 1.5-4 mmol/l to improve the aerobic capacity as measured by peak VO2 at exercise testing in GSD5 patients. Thirty molecularly defined MCA adults will be enrolled: to half of them randomly selected the dietary regimen will be prescribed, while subjects in the control group will follow their usual balanced diet. The evaluators will be blinded to the diet followed by the examined patient

DETAILED DESCRIPTION:
McArdle disease (myophosphorylase deficiency, glycogen storage disease type 5, GSD5, OMIM # 232600) is an inherited metabolic disorder of skeletal muscle. Affected patients suffer from genetically determined lack of the enzyme muscle glycogen phosphorylase, which is essential for glycogen metabolism. The condition is caused by homozygous or compound heterozygous mutations in the muscle glycogen phosphorylase gene (PYGM) located at chromosome 11q13. Many pathogenic mutations have been identified in the gene, which spans 20 exons, and many are population specific. The most common mutation in Northern Europe and North America is a nonsense mutation at Arg50stop (R50X) in exon 1 (previously referred to as R49X). A second frequent mutation in this population, and in Spanish patients, is Gly205Ser (G205S). McArdle disease is a rare disorder with an estimated incidence of 1:100,000.

Complete absence of muscle phosphorylase results in the inability to mobilize muscle glycogen stores, which are normally required as substrate for energy generation during anaerobic metabolism, which occurs during start of exercise and high-intensity efforts. In affected people, symptoms of fatigue and discomfort therefore occur within minutes of initiating any activity and during strenuous activity such as lifting heavy weights or walking uphill. If the activity is continued despite symptoms, a severe cramp (which is called a contracture in GSD5, because the muscle contraction is not caused by neural stimulation) occurs, which leads to muscle damage. If the damage is substantial, acute rhabdomyolysis may occur, which in turn can result in dark brown/black discoloration of urine (myoglobinuria). When rhabdomyolysis is severe, myoglobinuria can lead to acute renal failure, requiring treatment with dialysis.

In patients with GSD5, aerobic metabolism is limited and varies as a function of the availability of alternative fuels as a function of exercise and diet. The second wind phenomenon is illustrative. The phenomenon is characterized by the ability to increase work output after about 7-8 minutes of exercise. The second wind occurs as a consequence of increased availability and metabolism of alternative fuel substrates, preferentially glucose supplied from the liver, but also free fatty acids metabolized through oxidative phosphorylation and ketones produced by the liver. Despite these compensatory fuels, which can substitute for the absent glycogen breakdown in muscle, the capacity for oxidative phosphorylation is impaired in GSD5, because of an almost complete absence of pyruvate, a by-product of glycolysis.

Reduced oxidative phosphorylation in untrained patients with GSD5 in turn reduces oxygen consumption to approximately 35% of normal and there is a disproportionate increase in heart rate during exercise in patients with GSD5 compared with healthy controls. Thus, unconditioned people with GSD5 have very limited exercise capacity, which affects quality of life.

Most patients present in the second or third decade, although symptoms are often reported retrospectively from childhood. With advancing age a 20-25% proportion of patients develop fixed muscle weakness predominantly affecting the shoulder girdle. No clear cut genotype-phenotype correlation has been found to explain the clinical variation in severity observed even within families, but the influence of polymorphisms in other genes has been hypothesized.

Currently, there is no treatment for the condition. There have been a small number of randomized controlled treatment trials, however the largest number of participants in any previous study was 19.

Taking glucose prior to exercise alleviates muscle symptoms by inducing a 'second wind' at the onset of exercise, but has detrimental effects on weight if used too frequently. A Cochrane systematic review of training in GSD5 identified a few non-randomized trials of aerobic training or dietary manipulation either with supplements such as creatine or with shift towards lipid sources, which showed no harmful effect and suggest benefit over a number of months however long-tern results and confirmation on larger cohorts are warranted.

In spite of these indications, controlled training and dietary habits are seldom followed by patients, who experience significant limitations in activity of daily living and restriction in their participation.

A key limitation to exercise in GSD5 is the bottleneck in fuel flow through the Tri Carboxylic Acid (TCA) cycle, which is imposed by the minimal supply of glucosyl units from muscle glycogen and thus glycolytic flux to feed the TCA cycle.

Dietary manipulation has been identified since the eighties as a potential strategy to improve functioning in GSD5. In spite of initial indications for high protein regimens, later experimental comparison of high protein vs high carbohydrate diets indicated a superiority for the latter. Particular interest was also focussed on diets with predominant lipid energy source (ketogenic or low carbohydrate ketogenic LCKD) with the assumption that ketones are easily taken up by mitochondria and can substitute for the missing acyl-CoA moieties not provided by the staggering glycolysis blocked upstream for the inaccessibility of muscle glycogen. LCKD has a long history as a therapeutic strategy for several conditions (epilepsy, PDH defect, GLUT1 defect) with a good record of safety and efficacy and a poorer record of tolerability. Isolated experiences of LCKD have been carried out in GSD5 patients (maximum 4 patients) with promising results.

ELIGIBILITY:
Inclusion Criteria:

* molecularly defined Glycogen storage disease type 5, ability to perform a cycle ergometer exercise test

Exclusion Criteria:

* pregnancy,
* medical condition preventing a LCKD regimen (CPT2 or acyl-CoA deficiency, liver heart or kidney failure, unstable diabetes).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2019-03-25 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Change in maximal (peak) oxidative capacity (VO2max) | six months
  pre to post diet comparison of maximal O2 consumption attained during an incremental cycle ergometer test

SECONDARY OUTCOMES:
heart rate | six months
  change in the maximum heart rate during constant load cycling exercise (HR const)
maximal workload | six months
  change in maximal workload capacity (Wmax) at incremental cycle ergometer test
12 min walking test | six months
  the maximum walking distance in 12 minutes
Fatigue | six months
  self-rated severity of fatigue symptoms on a Fatigue Severity Scale (FSS). The FSS scoring is 1-7 on 9 averaged domains. 1 is minimal fatigue and 7 is maximal.
Short Form 36 (SF36) | six months
  the quality of life assessed using the 36-item Short Form Health Survey questionnaire (SF36). SF36 scoring is 0-100 with higher values indicating worse outcome
Disability | six months
  the functional disability assessed using the WHO Disability Assessment Schedule 2.0 (WHODAS 2.0). WHO-DAS 2.0 scoring is 0-100 with higher scores indicating worse outcome
exertion | six months
  the rate of Perceived Exertion during constant workload cycling (RPEconst) scored on a NRS scale 0-10 where 10 is maximum pain

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Martinuzzi, MD, PhD, Principal Investigator — IRCCS E Medea
Locations (1):
- IRCCS Medea, Conegliano, Treviso, Italy

IPD SHARING:
Plan to Share IPD: No
Anonymised data might be loaded on the European registry for muscle glycogenoses (EUROMAC)

REFERENCES:
- [Result] Quinlivan R, Martinuzzi A, Schoser B. Pharmacological and nutritional treatment for McArdle disease (Glycogen Storage Disease type V). Cochrane Database Syst Rev. 2014 Nov 12;2014(11):CD003458. doi: 10.1002/14651858.CD003458.pub5. PMID 25391139
- [Result] Busch V, Gempel K, Hack A, Muller K, Vorgerd M, Lochmuller H, Baumeister FA. Treatment of glycogenosis type V with ketogenic diet. Ann Neurol. 2005 Aug;58(2):341. doi: 10.1002/ana.20565. No abstract available. PMID 16049943
- [Result] Vorgerd M, Zange J. Treatment of glycogenosys type V (McArdle disease) with creatine and ketogenic diet with clinical scores and with 31P-MRS on working leg muscle. Acta Myol. 2007 Jul;26(1):61-3. PMID 17915573
- [Result] Cai QY, Zhou ZJ, Luo R, Gan J, Li SP, Mu DZ, Wan CM. Safety and tolerability of the ketogenic diet used for the treatment of refractory childhood epilepsy: a systematic review of published prospective studies. World J Pediatr. 2017 Dec;13(6):528-536. doi: 10.1007/s12519-017-0053-2. Epub 2017 Jul 12. PMID 28702868
- [Result] Muzykewicz DA, Lyczkowski DA, Memon N, Conant KD, Pfeifer HH, Thiele EA. Efficacy, safety, and tolerability of the low glycemic index treatment in pediatric epilepsy. Epilepsia. 2009 May;50(5):1118-26. doi: 10.1111/j.1528-1167.2008.01959.x. Epub 2009 Feb 12. PMID 19220406
- [Result] Roehl K, Sewak SL. Practice Paper of the Academy of Nutrition and Dietetics: Classic and Modified Ketogenic Diets for Treatment of Epilepsy. J Acad Nutr Diet. 2017 Aug;117(8):1279-1292. doi: 10.1016/j.jand.2017.06.006. PMID 28754198
- [Result] Paoli A, Bianco A, Damiani E, Bosco G. Ketogenic diet in neuromuscular and neurodegenerative diseases. Biomed Res Int. 2014;2014:474296. doi: 10.1155/2014/474296. Epub 2014 Jul 3. PMID 25101284
- [Derived] Martinuzzi A, Musumeci O, Stefan C, Vinante E, Ferrati A, Perillo C, Pesenti N, Toscano A. Low-carbohydrate ketogenic diet in Mc Ardle's disease: a single-blinded randomized controlled trial. J Neurol. 2025 Oct 15;272(10):698. doi: 10.1007/s00415-025-13405-5. PMID 41094169